CLINICAL TRIAL: NCT03133858
Title: Longitudinal Cohort Study - for the Treatment of Acute Postoperative Pain and Postoperative Delirium, Postoperative Cognitive Dysfunctions, and Chronic Pain.
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Head of the Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité - University Medicine Berlin, Charite University, Berlin, Germany
Other Study IDs: PainLong
Record Dates: First submitted 2017-04-24; First posted 2017-04-28 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Pain; Delirium; Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Pain; Delirium; Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adequate pain therapy is important aspect of perioperative care. Sequelae of inadequate pain management are patient dissatisfaction, post-operative nausea and vomiting (PONV), inadequate nutrition, lack of mobilization, and an increased risk for the development of further complications, such as postoperative delirium (POD). The use of patient-controlled analgesia (PCA) systems, which allow patients to self-administer analgesics, has improved pain management. Conventional i.v. PCA and the non-invasive administration of sufentanil sublingual tablets (ZALVISO®) are available. The aim of this investigation is to study patient controlled analgesia systems and to examine the incidence of POD, POCD and postoperative pain.

DETAILED DESCRIPTION:
There are strong evidence-based recommendations for an appropriate assessment and treatment of postoperative pain. Due to the complex and subjective nature of pain, an adequate pain therapy is an extremely challenging task, and the under- or overdosing of analgesics are common. An inadequate pain therapy leads to patient dissatisfaction, post-operative nausea and vomiting (PONV), inadequate nutrition, lack of mobilization, and an increased risk for the development of further complications, such as postoperative delirium (POD). Other long-term consequences of an insufficient postoperative analgesia include the chronification of pain and post-traumatic stress disorder (PTSD). Conversely, excessive opioid therapy may be associated with increased risk of POD. Subsequently, patients with POD have an increased risk for the consecutive development of postoperative cognitive dysfunction (POCD). The latter is marked by a progressive and permanent loss of cognitive abilities, which can ultimately lead to dementia. The use of patient-controlled analgesia (PCA) systems, which allow patients to self-administer analgesics, has been an improvement in the prevention of under- and overdosage of analgesics. Currently, there are two systems available: Conventional i.v. PCA with patients being dependent on an i.v. line and a PCA-pump and a patient-controlled, non-invasive administration of sufentanil sublingual tablets (ZALVISO®). The aim of this investigation is to study patient controlled analgesia systems and to examine the incidence of POD, POCD and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery with planned use of a patient-controlled analgesia system for postoperative pain therapy

Exclusion Criteria:

* Children (<18 years of age),
* Pregnancy and lactation
* Emergency surgery
* Accommodation in an institution due to an official or judicial order
* Participation in other clinical studies 30 days before study inclusion and during the study period
* Refusal of the patient
* Chronic opioid therapy > 3 months before surgery with an oral morphine sulfate equivalent >20mg/day
* Lacking willingness to save and hand out pseudonymized data within the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and female patients scheduled for elective surgical procedures in the fields of orthopedics, trauma surgery, gynecology, and urology, with planned patient-controlled analgesia used.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2021-11-28 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium (POD) | Until the 7th postoperative day
  The Nu-DESC (Nursing Delirium Screening Scale) and CAM-ICU (Confusion Assessment Method for the Intensive Care Unit) will be used as scoring systems to detect POD.
Incidence of postoperative cognitive deficit (POCD) | Up to one year
  The neuropsychological assessment will be performed at preoperative baseline until postoperative day 7, three-months and 1-year follow-up. In order to correct change in cognitive performance for practice effects, a group of non-surgical control subjects from the POCD Register (EA1/104/16) will also be evaluated with the cognitive test battery. The control subjects will be matched to the study group regarding health status, surgery and age.
Incidence of postoperative chronic pain | Up to one year
  The DSF (German pain questionnaire) and Ease of Care (EOC) questionnaire will be used to assess pain.

SECONDARY OUTCOMES:
Time until fully Mobilization (walking) after elective surgery (days) | Until the 7th postoperative day
Time to first oral nutritional intake (days) | Until the 7th postoperative day
Patient satisfaction | Until the 5th postoperative day
  Patient Global Assessment- patients overall satisfaction with procedure to reduce pain measured as 11-item likert scale
Postoperative complications | Until the 7th postoperative day
  Measurement includes adverse events of pain therapy
Pain intensity | Until the 7th postoperative day
  Numeric rating scale, mean of maximum and minimum- Course of patients pain intensity measured with 11-item likert scale
Amount of administered analgetics | Until the 7th postoperative day
Duration until discharge | Participants will be followed for the duration of hospital length of stay, an expected average of 3 weeks
Costs of pain therapy | Participants will be followed for the duration of hospital length of stay, an expected average of 3 weeks
Duration of pain therapy | Participants will be followed for the duration of hospital length of stay, an expected average of 3 weeks
Quality of life questionnaire | 3 months and 1 year after hospital discharge
  Quality of life will be measured with the EQ5D
Intensive care unit length of stay | Participants will be followed for the duration of intensive care stay, an expected average of 1 week
Mortality | Up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, MD, Prof., Study Director — Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité - University Medicine Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charité - University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borck M, Wandrey JD, Spies C, Tafelski S. Sublingual sufentanil after orthopaedic and abdominal surgery: long-term outcome and safety. Perioper Med (Lond). 2025 Feb 28;14(1):23. doi: 10.1186/s13741-025-00506-y. PMID 40022238